CLINICAL TRIAL: NCT01611571
Title: Combination Risedronate - Parathyroid Hormone Trial in Male Osteoporosis
Acronym: RPM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Alliance for Better Bone Health (Other)
Responsible Party: Principal Investigator, Marcella Walker, Irving Assistant Professor of Clinical Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAA4304
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Osteoporosis
Keywords: osteoporosis; male
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Risedronate Placebo Teriparatide (Active Comparator): Active Risedronate + Placebo Teriparatide for 18 months / Active Risedronate for 6 months
  Interventions: Drug: Risedronate; Drug: Placebo Teriparatide
- Active Risedronate Active Teriparatide (Active Comparator): Active Risedronate + Active Teriparatide for 18 months / Active Risedronate for 6 months
  Interventions: Drug: Risedronate; Drug: Teriparatide
- Placebo Risedronate Active Teriparatide (Active Comparator): Placebo Risedronate Active Teriparatide for 18 months / Active Risedronate for 6 months
  Interventions: Drug: Teriparatide; Drug: placebo Risedronate

INTERVENTIONS:
Drug: Risedronate — weekly risedronate
  Other Names: Actonel; Risedronic Acid
  Arms: Active Risedronate Active Teriparatide; Active Risedronate Placebo Teriparatide
Drug: Teriparatide — daily teriparatide
  Other Names: PTH1-34; Forteo
  Arms: Active Risedronate Active Teriparatide; Placebo Risedronate Active Teriparatide
Drug: Placebo Teriparatide — daily placebo of teriparatide
  Other Names: Teriparatide; PTH1-34; Forteo
  Arms: Active Risedronate Placebo Teriparatide
Drug: placebo Risedronate — weekly placebo of Risedronic Acid
  Other Names: Risedronate; Risedronic Acid
  Arms: Placebo Risedronate Active Teriparatide

SUMMARY:
The purpose of this study is to develop new treatment options for osteoporosis in men. The Investigators will study two medications and three treatment regimens. First, risedronate (FDA approved) will be studied as monotherapy. Second, the investigators will study injectable parathyroid hormone (PTH 134, teriparatide; FDA approved), as a therapy for male osteoporosis. PTH, a naturally occurring hormone produced by the parathyroid glands, is one of the most important regulators of bone metabolism. The drug being studied in this protocol, teriparatide, is the first aminoterminal 34 amino acids of the native 84amino acid peptide. Teriparatide contains all of the classical biological activities of native PTH. In studies of postmenopausal women, in a small study of 23 men with osteoporosis and a larger study of 437 men treatment with teriparatide led to significant increases in bone density. Although teriparatide and actonel are now approved for osteoporosis in men additional studies of these medications are needed in order to establish how best to use these drugs. This study is focused on an entirely new treatment approach, namely the combination of two medications for the treatment of osteoporosis risedronate with teriparatide to evaluate whether combination therapy is superior to therapy with either medication alone. This study is also designed to assess the extent to which risedronate maintains increases in bone density after a course of mono or combination therapy.

DETAILED DESCRIPTION:
Study Design:

This study involves a 24month commitment, constituting 12 visits as outlined below. The study coordinator will contact patients remotely by phone or email at the Month 9 visit, the Month 15, and the Month 21 visit so these do not require travel to Columbia University Medical Center.

This randomized, doubleblind study has two phases. The first 18month phase has 3 arms.

Patients will be randomized to receive either:

Risedronate / arm 1; 33% of total number of patients Teriparatide / arm 2; 33% of total population or, The combination of Teriparatide and Risedronate / arm 3; 33% of total population.

All patients will receive a daily subcutaneous injection with a small, 31 gauge needle (Teriparatide 20 ug or placebo vehicle), as well as a weekly pill (Risedronate 35 mg or placebo).

The second phase of the study will last for 6 months. During this time, patients will stop their daily injections but will continue taking weekly pills. These pills will contain Risedronate for all patients.

Thus, the second phase of the study, lasting 6 months, will have only one arm; that being, all participants will be on open label Risedronate for six months.

TOTAL: 90 men

Primary Endpoint: change in spine bone density in phase one of the study. The PRIMARY OUTCOME MEASURE in this study is the percentage change in lumbar spine bone density after 18 months of therapy comparing the three groups.

Power analysis was conducted based upon ascertaining significance of change of the first 18 months and the subsequent 6 months of the protocol. Based upon a 2-tailed test with an alpha of 0.05, the anticipated change in each of the three arms will be readily apparent at the lumbar spine with the "n" of 30 in each group.

Secondary Endpoint: change in LS bone density at 24 months, change in hip and radius bone density in phase one and phase two of the study, change in bone markers, morphometric vertebral fractures at 18 months.

VISIT ONE: Screening visit:

At this visit study staff will review the Consent Form (patient and person obtaining consent sign the consent form) and inclusion/exclusion criteria. They will collect demographic information, medical history, treatment history for patient's osteoporosis, and prior medication history.

Physical exam of the mouth, thyroid/neck, heart, lungs, abdomen, extremities, skin, mental status, sensory/motor status, lymph nodes, musculoskeletal, general appearance, height, weight, and blood pressure will be performed in order to identify any conditions which may exclude the potential participant from the study. This will be hereto forth referred to as "Physical Exam" Blood will be collected from the patient. A total of 2 tablespoons of blood by volume will be drawn from the patient to test for serum calcium, creatinine, parathyroid hormone, hepatic function, (Total Protein, Albumin, Globulin, A/G Ratio, Total Bilirubin, Direct Bilirubin, Alkaline Phosphatase, ALT, AST), and testosterone levels to determine the patient's eligibility for the study. Approximately 1.5 tablespoons of blood will be stored for research. The blood will be tested later for bone markers.

Duration: approximately 3 hours

VISIT TWO: Baseline/0 visit:

On this day patients begin their medications. Patients will learn how to administer injections (Teriparatide) and take the study pill (Risedronate) and will receive their first 6months worth of study supplies. The study drugs are managed by the Columbia University Research Pharmacy. The number of injection pens and the number of pills given to the patient will be recorded in case report forms. This will be hereto forth referred to as "Study Drug Supply/ ReSupply". In addition to the study drugs, the patients will be required to take a multivitamin with at least 400 IU of vitamin D and at least 500 mg of calcium each day. This is considered standard of care for people with osteoporosis. The patient will be asked if he/she experiences leg cramps, fatigue, depression, constipation, increased urination, back pain/kidney stones, local irritation/inflammation at the injection site or difficulty swallowing/esophageal ulcers, or dental problems such as the need to have a tooth pulled, implant placed or other dental procedure, nonhealing mouth sore. The patient can respond that these symptoms are absent, mild, moderate, or severe. This information is collected as a baseline for comparison to symptoms that may develop as a consequence of study medication usage.

This will be hereto forth referred to as "Adverse Events". Patients are asked about any changes in supplementary or prescription medications since the last visit. Patients are asked about any changes in treatments for conditions old or new since the last visit. Patients are asked if any medical conditions or events have occurred or significantly changed since the last visit. All information will be recorded in case report forms. This will be hereto forth referred to as "New Conditions/Con Meds".

Blood will be collected from the patient. A total of 2 tablespoons of blood by volume will be drawn from the patient. Approximately 0.5 tablespoons of blood will be used to test blood calcium and creatinine to monitor the safety of the patient. This will be hereto forth referred to as "Blood Calcium/Creatinine". Approximately 1.5 tablespoons of blood will be stored for research. The blood will be tested later for bone markers.

This will be hereto forth referred to as "Blood Storage." Urine will be collected from the patient. Urine will be collected over a 24hour period and stored for research and tested later for Calcium and Creatinine levels. This will be hereto forth referred to as "24 Hour Urine" Additionally, a spot urine sample will be collected from the patient at the visit. This will be stored for research and tested later for urine NTX. This will be hereto forth referred to as "Urine Storage" Xrays of the lumbar and thoracic spine (Lumbar and Thoracic AP and Lateral images) will be done to establish baseline fracture presence. This will be hereto forth referred to as "XRay".

Dual Xray Absorptiometry (DXA) will be performed to establish baseline bone density. This will be hereto forth referred to as "BMD" Duration: approximately 3 hours

VISIT THREE: Week 1:

Procedures that are repeated include Blood Calcium/Creatinine, Blood Storage, Urine Storage, 24 Hour Urine, Adverse Events, and New Conditions/Con Meds Duration: approximately 30 minutes

VISIT FOUR: Month 1:

Procedures that are repeated include Blood Storage, Urine Storage, Adverse Events, and New Conditions/Con Meds Duration: approximately 30 minutes

VISIT FIVE: Month 3:

Procedures that are repeated include Blood Calcium/Creatinine, Urine Storage, Adverse Events, and New Conditions/ Con Meds Duration: approximately 30 minutes

VISIT SIX: Month 6:

Procedures that are repeated include Physical Exam, Study Drug Supply/ ReSupply, Blood Calcium/Creatinine, Blood Storage, Urine Storage, BMD, Adverse Events, and New Conditions/Con Meds Duration: approximately 1.5 hours.

VISIT SEVEN: Month 9: phone visit:

Procedures that are repeated include Adverse Events, and New Conditions/Con Meds.

Duration: Approximately 15 minutes.

VISIT EIGHT: Month 12:

Procedures that are repeated include Study Drug Supply/ ReSupply, Blood Calcium/Creatinine, Blood Storage, Urine Storage, BMD, XRay, Adverse Events, and New Conditions/Con Meds Duration: approximately 2.5 hours.

VISIST NINE: Month 15: phone visit:

Procedures that are repeated include Adverse Events, and New Conditions/Con Meds Duration: Approximately 15 minutes.

VISIT TEN: Month 18:

Termination from phase 1 and entry into phase 2. Procedures that are repeated include Physical Exam, Blood Calcium/Creatinine, Blood Storage, Urine Storage, 24 Hour Urine, BMD, XRay, Adverse Events, and New Conditions/Con Meds. Study Drug Supply/ ReSupply will also occur. Of note, this will be Risedronate only, no more injectable medication). Patients therefore will only be given a supply of 6months worth of study pills.

Duration: approximately 2.5 hours

VISIT ELEVEN: Month 21: phone visit:

Procedures that are repeated include Adverse Events, and New Conditions/Con Meds Duration: Approximately 15 minutes.

VISIT TWELVE: Month 24: FINAL STUDY VISIT. Study physicians will discuss bone density results and recommend a course of poststudy treatment (if needed).

Procedures that are repeated include Physical Exam, Blood Calcium/Creatinine, Blood Storage, Urine Storage, 24 Hour Urine, BMD, XRay, Adverse Events, and New Conditions/Con Meds.

Termination from study occurs here. Duration: approximately 3.5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Males, ages 30-85 with osteoporosis.
2. Osteoporosis can be due to hypogonadism, past steroid use, or idiopathic.
3. Patients with hypogonadism can be included if their replacement dosage of testosterone has been stable for at least 18 months.
4. Bone mineral density must be 2 or more standard deviations below (T-score 2.0) the young adult peak for men at the lumbar spine, the hip or the radius.
5. Normal renal (glomerular filtration rate >= 60 ml/min) and liver (less than or equal to twice the normal limits for ALT and AST) function.

Exclusion Criteria:

1. Use of any specific osteoporosis drug in the previous 6 months.
2. Known or suspected metabolic bone diseases (such as renal osteodystrophy, osteomalacia) other than osteoporosis.
3. Preexisting hypercalcemia or an underlying hypercalcemic disorder, such as primary hyperparathyroidism.
4. Secondary hyperparathyroidism.
5. Paget's disease of bone or fibrous dysplasia. Teriparatide should not be given to patients with these conditions due to an increased risk of osteosarcoma.
6. Patients with any elevations of alkaline phosphatase that are secondary to bone disease, as such individuals may be at risk for osteosarcoma.
7. History or presence of any malignancy, except dermatological, but including melanoma. Known or suspected bone metastasis, or a history of skeletal malignancies.
8. Prior radiation therapy. Patients with prior radiation therapy should be excluded from treatment with teriparatide.
9. Any medical condition, which in the opinion of the investigator could preclude study participation, including but not limited to cardiovascular, gastric, renal and hepatic disorders, or abnormal PSA test. In particular, patients with active or recent (within the last 2 years) urolithiasis will be excluded.
10. History of previous major bowel surgery including bowel resection.
11. Oral use of systematic glucocorticoids for two or more weeks in the previous six months.
12. Parenteral use of systemic glucocorticoids on more than two occasions in the previous six months.
13. Use of anticonvulsant drugs.
14. History of uncontrolled diabetes mellitus (Patient with Type 2 diabetes who have HbA1C< 8 are permitted to be enrolled).
15. Hypercalciuria (> 4 mg/kg/day).
16. Impaired liver function (>twice the upper normal limits for ALT and AST).
17. Hyperadrenalism as assessed by physical examination.
18. Any other clinically significant laboratory abnormalities, which are deemed relevant to the design of the protocol.
19. Patients with known hypersensitivity to any of the test materials (teriparatide or risedronate) or related components (metacresol, mannitol, glacial acetic acid, sodium acetate).
20. Use of any investigational or unlicensed drug in the previous 30 days.
21. Patients who may be unreliable for the study, including those engaging in excessive alcohol consumption or drug abuse or patients who are unable to return for scheduled follow-up visits.
22. Patients who are unable or unwilling to comply fully with the protocol.
23. Inability to stand or sit upright for at least 30 minutes
24. Those with history of esophagitis, Barrett's esophagus, esophageal/peptic ulcers or esophageal motility disorders
25. Hypocalcaemia
26. Renal dysfunction (GFR <60)
27. Patients planning invasive dental work such as implants, extractions or procedures involving the jaw bone or patients with poor oral hygiene
28. Use of digitalis.
29. Patients with HIV/AIDS.

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Walker, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Harkness Pavilion, New York, New York, United States

REFERENCES:
- [Result] Walker MD, Cusano NE, Sliney J Jr, Romano M, Zhang C, McMahon DJ, Bilezikian JP. Combination therapy with risedronate and teriparatide in male osteoporosis. Endocrine. 2013 Aug;44(1):237-46. doi: 10.1007/s12020-012-9819-4. Epub 2012 Oct 26. PMID 23099796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: beginning 12/23/2003 and ending 11/2008 a total of 31 participants were enrolled in this study.
Groups:
- Active Risedronate + Active Teriparatide: Active Risedronate Active Teriparatide
  Risedronic acid & teriparatide : weekly risedronate daily teriparatide
- Active Risedronte + Placebo Teriparatide: Active Risedronte Placebo Teriparatide
  Risedronic acid : weekly risedronate daily teriparatide (placebo)
- Placebo Risedronate + Active Teriparatide, Active Risedronate: Placebo Risedronate Active Teriparatide for 18 months Active Risedronate for 6 months
  Teriparatide : weekly risedronate (placebo) 18 months daily teriparatide 18 months weekly risedronate 6 months
Period: Overall Study
Arm/Group | Active Risedronate + Active Teriparatide | Active Risedronte + Placebo Teriparatide | Placebo Risedronate + Active Teriparatide, Active Risedronate
Started | 11 | 10 | 10
Completed | 10 | 10 | 9
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Risedronate Active Teriparatide: Active Risedronate Active Teriparatide
  Risedronic acid & teriparatide : weekly risedronate daily teriparatide
- Active Risedronte Placebo Teriparatide: Active Risedronte Placebo Teriparatide
  Risedronic acid : weekly risedronate daily teriparatide (placebo)
- Placebo Risedronate Active Teriparatide, Active Risedronate: Placebo Risedronate Active Teriparatide for 18 months Active Risedronate for 6 months
  Teriparatide : weekly risedronate (placebo) 18 months daily teriparatide 18 months weekly risedronate 6 months
- Total: Total of all reporting groups
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide, Active Risedronate | Total
Number analyzed (Participants) | 11 | 10 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 31
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (4.9) | 54 (2) | 51.6 (3.9) | 51.6 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 10 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Spine Bone Density
Description: change in spine bone density at 18 months measured by DXA 18 and 24 months
Time Frame: 18 months
Measure: Least Squares Mean (Standard Deviation); unit: % change in LS BMD
Groups:
- Placebo Risedronate Active Teriparatide: Placebo Risedronate Active Teriparatide for 18 months Active Risedronate for 6 months
  Teriparatide : weekly risedronate (placebo) 18 months daily teriparatide 18 months weekly risedronate 6 months
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide
Number analyzed (Participants) | 10 | 10 | 9
% change in LS BMD | 6.95 (1.9) | 3.76 (1.8) | 5.68 (1.9)

2. Secondary Outcome: Change in Hip Bone Density
Description: change in hip bone density measured by DXA
Time Frame: baseline and 18 months
Measure: Mean (Standard Deviation); unit: % change in TH BMD
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide
Number analyzed (Participants) | 10 | 10 | 9
% change in TH BMD | 3.86 (1.1) | 0.82 (0.95) | 0.29 (0.95)

3. Secondary Outcome: Change in Forearm Bone Density
Description: change in 1/3 radius of forearm bone density as measured by DXA
Time Frame: baseline and 18 months
Measure: Mean (Standard Deviation); unit: % change in 1/3 Radius BMD
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide
Number analyzed (Participants) | 10 | 10 | 9
% change in 1/3 Radius BMD | 1.6 (0.6) | 0.11 (0.77) | 0.02 (0.77)

4. Secondary Outcome: New Morphometric Vertebral Fractures
Description: counting the total new morphometric vertebral fractures as determined by x-ray from baseline through end of study
Time Frame: baseline through 18 months
Measure: Number; unit: vertebral fracture
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide
Number analyzed (Participants) | 10 | 10 | 9
vertebral fracture | 1 | 1 | 0

5. Secondary Outcome: Change in FN BMD at 18 Months
Description: Change in the Femoral Neck BMD at 18 month
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: % change in TH BMD
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide
Number analyzed (Participants) | 10 | 10 | 9
% change in TH BMD | 8.45 (1.8) | 0.5 (1.7) | 3.89 (1.7)

ADVERSE EVENTS:
Time Frame: each participant was enrolled for a total of 24 months and adverse events were collected throughout the entirety of their participation.
Arm/Group | Active Risedronate Active Teriparatide | Active Risedronte Placebo Teriparatide | Placebo Risedronate Active Teriparatide, Active Risedronate
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Risedronate Active Teriparatide (N=10) | Active Risedronte Placebo Teriparatide (N=10) | Placebo Risedronate Active Teriparatide, Active Risedronate (N=9)
Fracture, patella (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — fracture of the left patella. This fracture not deemed to be a fragility fracture or in any way related to study drug or participation in the study.
Fracture, vertebral (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) — new vertebral fracture
Fatigue (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (4) | 1 (3) | 0 (0)
Injection Site Irritation (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (6) | 1 (1)
Difficulty Swallowing (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Leg Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) — participants experienced either leg cramping for the first time, or worsening of existing leg cramping
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No